CLINICAL TRIAL: NCT03554499
Title: Bichectomy: Hydrodissection Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Dr. Ruben Leñero (Other)
Responsible Party: Principal Investigator, LUIS VALENCIA, PLASTIC SURGERY RESIDENT, Hospital General Dr. Ruben Leñero
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2050100617
Record Dates: First submitted 2018-05-09; First posted 2018-06-13 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Aging
Keywords: Facial aging; Buccal fat pad

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrodissection (Experimental): Bichectomy with hydrodissection = infiltration of 15ml per side of a special solution (250ml of saline 0.9% + 1mg of epinephrine + 20ml of 2% Lidocaine, equivalent to 0.0555mg of epinephrine and 22.2mg of Lidocaine per side), prior to the incision with the following distribution: 1ml in the form of a wheal in the oral mucosa with a 22G needle 1cm behind the Stenon canal opening that corresponds to the incision site and 14 ml on the virtual space where the buccal fat pad is located.
  Interventions: Procedure: Bichectomy with hydrodissection
- Control (Active Comparator): Bichectomy without hydrodissection = infiltration with 3ml per side of 2% Lidocaine with 1: 200,000 epinephrine ( equivalent to 0.015mg of epinephrine and 60mg of Lidocaine per side) at the operative site.
  Interventions: Procedure: Bichectomy

INTERVENTIONS:
Procedure: Bichectomy with hydrodissection — Intraoral removal of buccal fat pads using hydrodissection technique
  Other Names: Bichatectomy
  Arms: Hydrodissection
Procedure: Bichectomy — Intraoral removal of buccal fat pads using conventional technique
  Other Names: Bichatectomy
  Arms: Control

SUMMARY:
Buccal Fat Pad provides volume to the middle third of the face and occasionally may cause deepening of the nasolabial fold and relaxation of the mimetic muscles, both associated with aging. Bichectomy is the surgical procedure in which the buccal fat pad is remove in order to achieve a youthful and aesthetic appearance, getting harmony in facial contour. The purpose of this study was to compare the usual technique with an alternative method, using hydrodissection to facilitate the dissection of the Buccal Fat Pad making this procedure safer, efficient and more pleasant for the patient.

DETAILED DESCRIPTION:
This is a randomized controlled trial primarily designed to compare an alternative method for Bichectomy using hydrodissection. All procedures were performed by the same surgeon using the same technique, the only difference was the infiltration methods.

1. Two groups were assigned:

   * Group A - Bichectomy with hydrodissection = infiltration of 15ml per side of a special solution (250ml of saline 0.9% + 1mg of epinephrine + 20ml of 2% Lidocaine, equivalent to 0.0555mg of epinephrine and 22.2mg of Lidocaine per side), prior to the incision with the following distribution: 1ml in the form of a wheal in the oral mucosa with a 22G needle 1cm behind the Stenon canal opening that corresponds to the incision site and 14 ml on the virtual space where the buccal fat pad is located, which is immediately identified after penetrating the fascia of the buccinator muscle where you can feel a difference in resistance.
   * Group B - Bichectomy without hydrodissection = infiltration with 3ml per side of 2% Lidocaine with 1: 200,000 epinephrine ( equivalent to 0.015mg of epinephrine and 60mg of Lidocaine per side) at the operative site.
2. Inclusion criteria : Adult patients older than 18 years old with a round face and prominent cheeks undergoing bichectomy to improve aesthetic facial contour during the period April 2016 and October 2017.
3. Exclusion criteria : Patients with previous facial procedures, malar hypoplasia, obesity, metabolic diseases, coagulopathies or neuropathy diagnosis confirmed by a neurologist.
4. Patient Sample : Total of 54 patients were included.
5. Surgical technique: patient lay down at 30º angle, a 0.5cm incision of the mucosa with a 15 blade in a horizontal fashion placed 1cm posterior to stenon canal opening, then a Kelly clamp is introduce pushing towards the ear lobe until a resistance is passed which corresponds to the buccinator fascia, the Kelly clamp is opened following the buccinators muscle fibers direction and the fat pad is immediately identified, extracted, and leaving the wound open for closure by second intension.
6. Variables analyzed:

   6.1) Transoperative pain - Patients were provided with a validated visual analogue scale (VAS) for pain and asked to rate their pain in a range of 0-10

   6.2) Postoperative pain at 2 hours - Patients were provided with a validated visual analogue scale (VAS) for pain and asked to rate their pain in a range of 0-10.

   6.3) Maximum pain in first 72 hours postoperative - Patients were provided with a validated visual analogue scale (VAS) for pain and asked to rate their pain in a range of 0-10.

   6.4) Procedure time - surgical time was quantified with a digital chronometer (IPhone 5s) managed by an independent operator, from the initial incision to the time of extraction for both fat pads.

   6.5) Bleeding - was recorded by measuring total number of soaked gauze with each piece of gauze holding 5cc of blood.

   6.6) Complications - complications were collected prospectively, defined as being within the first 90 postoperative days.
7. Postoperative care was standardized and patients were followed up for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years with a round face and prominent cheeks undergoing bichectomy to improve aesthetic facial contours

Exclusion Criteria:

* Patients with previous facial procedures, malar hypoplasia, obesity, metabolic diseases, coagulopathies or neuropathy diagnosis confirmed by a neurologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04-02 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
TRANSOPERATIVE PAIN | 1 DAY
  INVESTIGATORS ASK THE PATIENTS TO RATE THEIR PAIN PERCEPTION USING THE VISUAL ANALOG SCALE FOR PAIN (VAS PAIN), USING A NUMERICAL RATING SCALE FROM 0 (NO PAIN) - 10 (SEVER PAIN)
2 HOURS POSTOPERATIVE PAIN | 1 DAY
  INVESTIGATORS ASK THE PATIENTS TO RATE THEIR PAIN PERCEPTION USING THE VISUAL ANALOG SCALE FOR PAIN (VAS PAIN), USING A NUMERICAL RATING SCALE FROM 0 (NO PAIN) - 10 (SEVER PAIN)
MAXIMUM PAIN IN FIRST 72 HOURS POSTOPERATIVE. | 3 DAYS
  INVESTIGATORS ASK THE PATIENTS TO RATE THEIR PAIN PERCEPTION USING THE VISUAL ANALOG SCALE FOR PAIN (VAS PAIN), USING A NUMERICAL RATING SCALE FROM 0 (NO PAIN) - 10 (SEVER PAIN)

SECONDARY OUTCOMES:
SURGICAL TIME | DURING PROCEDURE
  PROCEDURE TIME IN MINUTES SINCE THE FIRST INCISION TO THE END OF THE PROCEDURE
BLEEDING | DURING PROCEDURE
  1GAUZE = 5ML
COMPLICATIONS | 90 DAYS
  COMPLICIATIONS PRESENTED AFTER PROCEDURE

REFERENCES:
- [Background] Jackson IT. Buccal fat pad removal. Aesthet Surg J. 2003 Nov-Dec;23(6):484-5. doi: 10.1016/j.asj.2003.08.005. PMID 19336124
- [Background] Matarasso A. Buccal fat pad excision: aesthetic improvement of the midface. Ann Plast Surg. 1991 May;26(5):413-8. doi: 10.1097/00000637-199105000-00001. PMID 1952712
- [Background] Khiabani K, Keyhan SO, Varedi P, Hemmat S, Razmdideh R, Hoseini E. Buccal fat pad lifting: an alternative open technique for malar augmentation. J Oral Maxillofac Surg. 2014 Feb;72(2):403.e1-15. doi: 10.1016/j.joms.2013.10.002. Epub 2013 Oct 16. PMID 24438602
- [Background] Eber Luis de L S. Bichectomy or Bichatectomy - A Small and Simple Intraoral Surgical Procedure with Great Facial Results. Adv Dent & Oral Health. 2015; 1(1): 555555. doi: 10.19080/ADOH.2015.01.555555
- [Background] Xu J, Yu Y. A modified surgical method of lower-face recontouring. Aesthetic Plast Surg. 2013 Apr;37(2):216-21. doi: 10.1007/s00266-013-0080-x. Epub 2013 Feb 16. PMID 23417575
- [Background] Yousuf S, Tubbs RS, Wartmann CT, Kapos T, Cohen-Gadol AA, Loukas M. A review of the gross anatomy, functions, pathology, and clinical uses of the buccal fat pad. Surg Radiol Anat. 2010 Jun;32(5):427-36. doi: 10.1007/s00276-009-0596-6. Epub 2009 Nov 25. PMID 19937328
- [Background] Quispe GD, Lupa C. Cirugía estética de mejillas. Rev Act Clin Med 2014;48:2538-2541. ISSN 2304-3768.
- [Background] Hasse FM, Lemperle G. Resection and augmentation of Bichat´s fat pad in facial contouring. Eur J Plast Surg. 1994;17:239-242. doi: 10.1007/BF00208838
- [Background] Bayter JE. Manejo de líquidos, lidocaína y epinefrina en liposucción. Rev Colomb Anestesiol. 2015;43(1):95-100. doi:10.1016/j.rca.2014.09.007
- [Background] Stuzin JM, Wagstrom L, Kawamoto HK, Baker TJ, Wolfe SA. The anatomy and clinical applications of the buccal fat pad. Plast Reconstr Surg. 1990 Jan;85(1):29-37. doi: 10.1097/00006534-199001000-00006. PMID 2293733
- [Background] Matarasso A. Managing the buccal fat pad. Aesthet Surg J. 2006 May-Jun;26(3):330-6. doi: 10.1016/j.asj.2006.03.009. PMID 19338917